CLINICAL TRIAL: NCT01640119
Title: A Prospective, Controlled, Randomized, Multicentric Study: Correction of Metabolic Acidosis With Use of Bicarbonate in Chronic Renal Insufficiency (CKD3b-4)
Brief Title: Correction of Metabolic Acidosis in End Stage Renal Disease (ESRD)
Acronym: UBI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Sanitaria ASL Avellino 2 (Other)
Responsible Party: Principal Investigator, Dr Biagio Di Iorio, Principal Investigator, Azienda Sanitaria ASL Avellino 2
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: aslav2
Record Dates: First submitted 2012-06-28; First posted 2012-07-13 (Estimated); Last update posted 2014-09-19 (Estimated); Status verified 2014-09

CONDITIONS: Metabolic Acidosis
Keywords: metabolic acidosis; renal death
MeSH Terms: conditions — Acidosis | interventions — Bicarbonates; Alkalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- no intervention (Placebo Comparator)
- Bicarbonate (Experimental)
  Interventions: Dietary Supplement: Bicarbonate

INTERVENTIONS:
Dietary Supplement: Bicarbonate — bicarbonate administration
  Other Names: Alkali
  Arms: Bicarbonate

SUMMARY:
The investigators want to evaluate whether an original action based on the administration of alkali (mainly sodium bicarbonate) is able to significantly modify renal death and to reduce mortality due to cardiovascular events.

Methods: This is a proposal of Multicentric, prospective, cohort, randomized, open-label and controlled study.

The investigators will Randomize 728 patients with Chronic Kidney Disease(CKD) stage 3b (CKD-3b) and CKD stage 4: 364 of these patients will be included in the study group called Bicarbonate Group (Bic), in which levels of bicarbonate should be kept > 24 mEq/l; the other 364 patients will included in the Usual Treatment Group (no-Bic).

Results: The aim of the Research Protocol is to demonstrate if that the optimal correction of uremic acidosis (with administration of sodium bicarbonate or of any other alkalinizing agent, e.g. sodium citrate) reduces renal and cardiovascular mortality.

Conclusions. In conclusion the Work Group of the Conservative Therapy for Chronic Renal Insufficiency proposes this cohort, randomized, controlled, prospective, multicentric study to evaluate the effects of correction of acidosis on the progression of the kidney disease considered as renal death in End-Stage Renal Disease (ESRD) patients.

DETAILED DESCRIPTION:
Rationale:

Chronic Kidney Disease (CKD) is associated with a high incidence of morbility and mortality.

In this regard, the National Health and Nutrition Examination Survey (NANHES) shows that 19% of the uremic population presents metabolic acidosis (CKD stage 4). This high prevalence and the low costs of the correction by bicarbonate pave the way for a potential and interesting research activity.

In fact, a Cochrane Collaboration review reports that there is no evidence for correction of acidosis by sodium bicarbonate in pre-End-Stage Renal Disease) (ESRD) patients, and concludes that randomized controlled trials (RCTs) are necessary to evaluate the benefits and harms of correcting metabolic acidosis in pre-ESRD patients.

During the same year, 2009, another RCT appears in the scientific literature showing that the administration of sodium bicarbonate, and the consequent correction of acidosis, slows the progression of CKD and improves the nutritional status in ESRD patients stages 4-5. This study was randomized, prospective, open-label, monocentric, and was conducted on 134 patients.

It is well known that acidosis stimulates proteic catabolism, accelerates branched-chain amino acid oxidation and reduces the synthesis of visceral proteins. The beneficial effects of bicarbonate in experimental models in rats and the effects of correcting acidosis on the nutritional status are also known.

Less information is available on the possibility that correcting acidosis in pre-ESRD patients slows renal death and improves outcomes also in the future, on dialysis.

The above cited study of Brito and Ashurst highlights that bicarbonate supplementation (that causes the blood value to increase from 20 to 22 mmol/L) slows the rate of progression of CKD and betters the nutritional status of patients.

Moreover, very recently the author Menon has demonstrated that low levels of serum bicarbonate increase the risk of outcomes, e.g. renal death and mortality.

Finally, an article recently published on Kidney International has put in evidence the pathogenetic factors, e.g. endothelin and hyperaldosteronism, which were caused to worsen renal function in rats by the presence of metabolic acidosis.

In response to this article, an editorial by the authors Sahni, Rosa and Batlle D. has been published on the same issue of Kidney International with the following statement:

"There is increasing evidence that alkali therapy can retard progression of chronic kidney disease (CKD). We summarize recent studies and discuss a mechanism whereby alkali therapy may neutralize acid production associated with typical Western diets, which generate acid. We emphasize the rationale for using alkali therapy early in the course of CKD, even in the absence of overt metabolic acidosis, and we urge the pharmaceutical industry to develop palatable alkali- containing solutions."

Proposal for the study For the reasons explained above, the Work Group of the Conservative Therapy for Chronic Renal Insufficiency proposes this cohort, randomized, controlled, prospective, multicentric study to evaluate the effects of correction of acidosis on the progression of the kidney disease considered as renal death in ESRD patients.

Objectives:

Main objective:

1. To evaluate whether an original action based on the administration of alkali (mainly sodium bicarbonate) is able to significantly modify progression of renal disease, and renal death, and to reduce mortality due to cardiovascular events.
2. To verify if bicarbonate therapy modify progression of renal disease, and renal death, and to reduce mortality due to cardiovascular events in APKD patients.
3. To verify if bicarbonate therapy modify progression of renal disease, and renal death, and to reduce mortality due to cardiovascular events in dianetic patients.

Other objectives:

To evaluate if nutritional parameters improve during the period of study; To evaluate blood pressure (as absolute value and as increase in antihypertensive drugs); To evaluate how the correction of acidosis influences bone turnover (vascular calcifications); To evaluate changes in calcium and phosphorus metabolism.

Study design Multicentric, prospective, cohort, randomized and controlled study.

Randomize 728 patients with CKD-3b and CKD-4: 364 of these patients will be included in the study group called Bicarbonate Group (Bic), in which levels of bicarbonate should be kept > 24 mEq/l; the other 364 patients will included in the Usual Treatment Group (no-Bic).

Run-in period with one visit per month for 3 months, followed by a 36-month study period.

The investigated patients must be randomized by sex, diabetes and level of renal function (measured Clearance of Creatinine between 60 and 30 ml/min, between 30 and 15, <15 on pre-dialysis) and all the requirements for a Best Practice Treatment (BPT) must be applied:

* For anemia (Hb 11-12 g/dl; TSAT > 20 %),
* For arterial hypertension (systolic blood pressure (SBP) <130 mmHg; diastolic blood pressure (DBP) < 90 mm g),
* For hyperlipidemia (low-density (LDL) cholesterol <100),
* For osteodystrophy (phosphatemia 2.7-4.6 mg/dl; calcemia 8.4-10.2 mg/dl; in CKD-3: parathyroid hormone (PTH) 35-70 pg/ml; in CKD-4: PTH 70-110 pg/ml; 25(OH) vitamin D > 30 nmol/l).

(Failure to reach the BPT target will not cause exclusion as the centralized randomization will probably be the reason for the enrollment of patients who have the same clinical characteristics and the same treatments during the follow-up period).

Randomization will be centralized and patients will be randomized on the basis of sex, age, diabetes, levels of renal function (measured).

All patients will be provided with a nutritional and diet counseling consisting of a low protein, phosphorus and sodium diet.

Duration of the study:

3 years.

Primary endpoints

* Doubling of Creatinine

  . Beginning of dialysis
* All-cause mortality

Study Power

To determine the sample size was used EAST software version 3.1 and considered the following assumptions:

1. alfa 0.05;
2. power 0.90;
3. treatment/untreatment 1;
4. lost to follow-up 10 %;
5. Two-tailed statistical test with type I error of 5%.
6. Statistical power of the test equal to 80%.

Therefore, it was determined:

* Number of events required 194.
* Number of subjects needed 728
* Study duration 36 months.

Parameters measured every 3-6 months:

Bicarbonate levels blood albumin levels, fetuin-A, C-reactive protein blood levels of sodium, potassium, bicarbonate, chloride, blood levels of homocysteine, lipid profile blood levels of calcium, phosphorus, PTH, alkaline phosphatase, bone turnover markers blood levels of creatinine, plasma urea, blood count 24h urinary urea excretion, 24h urinary sodium excretion, 24h urinary protein excretion, 24 urinary creatinine excretion bioelectrical impedance assessment (BIA), body weight, blood pressure, Lateral abdominal X-ray for vascular calcification.

Use of anti-hypertensive drugs and diuretics.

Administration of bicarbonates:

The molecular weight of sodium bicarbonate is 84.01. Each gram of substance therefore contains 11.9 mmol, so initially as much as 3-4 grams can be administered, subsequently it has to be adjusted according to the blood level of bicarbonate.

Evaluations should be made on a bimonthly basis in order to adjust the administration of bicarbonate according to blood levels of bicarbonate (target values >24 e <28 mEq/L).

Bicarbonate administration should be suspended if blood bicarbonate levels are > 28 mEq/L.

For ethical reasons, partial correction of acidosis is allowed (up to 22 mEq/L) for blood bicarbonate levels lower than 18 mEq/L.

The aim of the study is to demonstrate that the optimal correction of uremic acidosis (with administration of sodium bicarbonate or of any other alkalinizing agent, e.g. sodium citrate) reduces renal and cardiovascular mortality.

Prerequisites of the study:

a) to expose the patient to low risks of unfavourable events, c) patients will be asked for a little but constant effort with some modifications in their life style, d) costs should be low for the family and for the institution where the patient is treated. No specific equipment and competences are required, so that the study can be easily performed in any Nephrology Division.

------------------------- Ethical aspects The physician will describe the study in detail and will read all information regarding the study to the patient so that he/she will have the opportunity to ask for any further clarification.

Thereafter, the patients will be provided with the Informed Consent, which he/she should sign after reading it throughout (see attachments). Patient's data will be recorded, processed and stored in complete accordance with the data protection laws, in order to safeguard the safety and privacy of data; if included in publications and/or presented at conferences, data will undergo a statical process and will be kept anonymous.

Statistics Methods of descriptive and distribution statistics together with parametric and non-parametric tests will be applied. Linear correlation or the Spearman test will be used to analyse the relationship between two variables considered simultaneously; the relationship among more variables will be analysed with multiple regression (linear or logistic).

ELIGIBILITY:
Inclusion Criteria:

* End stage renal disease

Exclusion Criteria:

* Neoplastic diseases

  * Autoimmune diseases
  * Decompensation class III-IV
  * Uncontrollable hypertension
  * Amputation of the limbs
  * Previous ictus cerebri
  * Neobladder, ureterosigmoidostomy
  * Sever acidosis with bicarbonate < 18 mEq/l
  * Use of calcium carbonate (relative exclusion factor: patients who used to take this drug and suspended it before the beginning of the 3-month run-in period can be included in the study).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 728 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
doubling of creatinine | 36 months
  the primary outcome will be reached when the seric creatinine level (mg/dl) will double compared to the basal value.

SECONDARY OUTCOMES:
all-cause death | 36 month
  all-cause death of patients
start of renal replacement therapy | 36 month
  start of dialysis (peritoneal dialysis or hemodialysis)

CONTACTS AND LOCATIONS:
Overall Officials: Biagio Di Iorio, MD, PhD, Principal Investigator — Azienda Sanitaria ASL Avellino 2
Locations (2):
- Italy (2):
  - UOC di Nefrologia, Solofra, Avellino
  - UOC do Nefrologia, Solofra, Avellino

REFERENCES:
- [Background] 1.Eustace JA, et al. Prevalence of acidosis and inflammation and their association with low serum albumin in chronic kidney disease. Kidney Int. 2004 ;65:1031-40. 2.Ballmer PE, et al: Chronic metabolic acidosis decreases albumin synthesis and induces negative nitrogen balance in humans. J Clin Invest 1995;95:39-40 3.Chiu YW, et al: Correction of metabolic acidosis to ameliorate wasting in chronic kidney disease: goals and startegies. Sem Nephrol 2009;29:67-74 4.Bommer J, et al: association of predialysis serum bicarbonate levels with risk of mortality and hospitalization in the DOPPS. Am J Kidney Disease 2004;44:661-671 5.Wu DY, et al: Association between serum bicarbonate and death in hemodialysis patients: is it better to be acidosis or alkalotic? Clin J Am Soc Nephrol 2006;1:70-78 6.Kraut JA, Madias NE. Metabolic acidosis: pathophysiology, diagnosis and management. Nat Rev Nephrol. 2010;6:274-85. 7.Roderick P, et al. Correction of chronic metabolic acidosis for chronic kidney disease patients. Cochrane Database Syst Rev. 2007; Jan 24(1):CD001890. 8.de Brito-Ashurst I, et al: Bicarbonate supplementation slows progression of CKD and improves nutritional status. J Am Soc Nephrol 2009;20:2075-2084 9.Menon V, et al: Serum bicarbonate and long-term outcomes in CKD. Am J Kidney Disease 2010; 56:907-14 10.Wesson DE, Simoni J: Acid retention during kidney failure induces endothelin and aldosterone production which lead to progressive GFR decline, a situation ameliorated by alkali diet. Kidney Int 2010;78 1128-1135
- [Derived] Di Iorio BR, Bellasi A, Raphael KL, Santoro D, Aucella F, Garofano L, Ceccarelli M, Di Lullo L, Capolongo G, Di Iorio M, Guastaferro P, Capasso G; UBI Study Group. Treatment of metabolic acidosis with sodium bicarbonate delays progression of chronic kidney disease: the UBI Study. J Nephrol. 2019 Dec;32(6):989-1001. doi: 10.1007/s40620-019-00656-5. Epub 2019 Oct 9. PMID 31598912
- [Derived] Bellasi A, Di Micco L, Santoro D, Marzocco S, De Simone E, Cozzolino M, Di Lullo L, Guastaferro P, Di Iorio B; UBI study investigators. Correction of metabolic acidosis improves insulin resistance in chronic kidney disease. BMC Nephrol. 2016 Oct 22;17(1):158. doi: 10.1186/s12882-016-0372-x. PMID 27770799